CLINICAL TRIAL: NCT05771207
Title: Effects of Soy Protein and Whey Protein on Muscle, Gut Microbiota and Clinical Outcome in Patients With Lung Cancer-related Sarcopenia（LCRS）: a Randomized, Double-blind, Controlled Clinical Study
Brief Title: Effects of Protein on Muscle, Gut Microbiota and Clinical Outcome in Patients With Lung Cancer-related Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yu Kang, MD, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: protein-cancer-sarcopenia2023
Record Dates: First submitted 2023-02-23; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer; Sarcopenia
Keywords: soy protein; whey protein; lung cancer related sarcopenia
MeSH Terms: conditions — Lung Neoplasms; Sarcopenia | interventions — Soybean Proteins; Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- soy protein intervention (Experimental): This group received dietary guidance and soy protein intervention for 3 months
  Interventions: Dietary Supplement: soy protein
- whey protein intervention (Experimental): This group received dietary guidance and whey protein intervention for 3 months
  Interventions: Dietary Supplement: whey protein
- control (Placebo Comparator): This group received dietary guidance and ｍltodextrin for 3 months
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: soy protein — The intervention is made up of soy protein supplements (30g/d) and dietary pattern modification.
  Arms: soy protein intervention
Dietary Supplement: whey protein — The intervention is made up of whey protein supplements (30g/d) and dietary pattern modification.
  Arms: whey protein intervention
Dietary Supplement: placebo — The intervention is made up of maltodextrin (30g/d) and dietary pattern modification.
  Arms: control

SUMMARY:
Sarcopenia is common in lung cancer patients. It is one of the significant factors affecting the overall survival, radiotherapy and chemotherapy efficacy, and quality of life of patients with lung cancer. Previous studies have shown that increased protein intake can stimulate postprandial muscle synthesis, and improve muscle mass, strength, function, and overall survival. However, most previous studies have focused on the intervention of whey protein, while the protective effect of soybean protein on lung cancer-related sarcopenia (LCRS) has not yet been fully explored and reached an agreement.

So, this study aims to explore the effects of soy and whey protein on muscle, gut microbiota, and clinical outcomes among patients with lung cancer-related sarcopenia, to provide a reference for further nutrition treatment.

DETAILED DESCRIPTION:
This study will last 6 months. For the duration of the study, an anticipated total of 90 participants will be randomly assigned to receive either a 30-gram protein supplement or a placebo daily. There will be a total of 5 study visits, and dietary records, questionnaires, blood and stool collection, and functional testing will occur at all study visits. Intention-to-treat analysis (ITT) and per-protocol analysis (PP) will be conducted in statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* age>=18years old
* Patients with lung cancer and sarcopenia
* ECOG<=2
* Patients are able to provide written informed consent.

Exclusion Criteria:

* People who are allergic to soy protein and whey protein.
* Participants received any drugs or supplements known to influence effcet size, such as protein powder, anabolic steroids, or glucorticosteroid before the 3 months preceding the study.
* Participants with gastrointestinal bleeding, enterotomy or gastric bypass surgery before the 3 months preceding the study.
* Concurrent severe cardiac disease, liver and renal failure, which may significantly interfere with study compliance.
* Participants with electronic or mental device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Appendicular skeletal muscle mass index at 3 months | 3 months
  Defined as muscle mass (Unit: kg/m2)

SECONDARY OUTCOMES:
Change from Baseline Hand grip at 3 months | 3 months
  Defined as muscle strength (Unit: kg)
Change from Baseline physical performance Baseline at 3 months | 3 months
  Measured by Short Physical Performance Battery (0-12) with higher scores meaning better physical performance.
Change from Baseline Physical function at 3 months | 3 months
  Measured by FRAIL scale (0-5) with higher scores meaning better physical function.
Change from Baseline Quality of life questionnaire at 3 months | 3 months
  Measured by EuroQol- 5 Dimension scale (0-5) with higher scores meaning better Quality of life.
Change from Baseline gut microbiota composition at 3 months | 3 months
  The stool samples of participants before and after intervention were collected and analized by 16S rRNA.
Number of patients with good Chemotherapy Tolerance | 3 months
  Completing initially planned chemotherapy course is defined as good tolerance; dose adjustment, delayed completion or interruption of treatment are considered as poor tolerance.
Incidence of Chemotherapy toxicity | 3 months
  Measured after initiation of chemotherapy using the WHO Toxicity Grades (gradeI-IV) with higher grades neaning severer chemotheraphy toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No